CLINICAL TRIAL: NCT04362722
Title: A Phase II Study of Intratumoral Administration of L19IL2/L19TNF in Non-melanoma Skin Cancer Patients With Presence of Injectable Lesions
Brief Title: Intratumoral Administration of Daromun in Non-melanoma Skin Cancer Patients
Acronym: DUNCAN
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Philogen S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PH-L19IL2TNFNMSC-04/19
Record Dates: First submitted 2020-04-17; First posted 2020-04-27 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Carcinoma, Basal Cell; Carcinoma, Cutaneous Squamous Cell
MeSH Terms: conditions — Carcinoma, Basal Cell; Carcinoma | interventions — daromun

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Experimental): 40 patients will be enrolled and treated with a mixture of 6.5 Mio IU (~1.08 mg) L19IL2 and 200 µg L19TNF once weekly for 4 consecutive weeks. The dose will be distributed among the lesions via multiple intralesional injections.
  New lesions occurring during the treatment phase will also be treated as described but the treatment period for new lesions will not be extended beyond the previously defined 4 weeks treatment period with clock-start at the time of the first intralesional L19IL2/L19TNF injection.
  After the Tumor Assessment/Safety visit, patients may receive surgery in a curative intention within 6 weeks, in order to assess the pathological response with estimation of percent of residual viable tumor cells.
  Interventions: Drug: L19IL2 +L19TNF

INTERVENTIONS:
Drug: L19IL2 +L19TNF — Single or multiple intratumoral administration of a mixture of L19IL2 and L19TNF will be performed once weekly for up to 4 weeks into all injectable lesions present at the beginning of treatment or appearing during treatment phase The dose will be constituted by 6.5 Mio IU L19IL2 (~1.08 mg) and 200 µg L19TNF.
  Other Names: bifikafusp alfa + onfekafusp alfa

SUMMARY:
This clinical phase II study is designed to investigate the efficacy of intratumorally administered L19IL2/L19TNF in patients with injectable lesions of BCC or cSCC. Favorable tumor responses following intralesional treatment with L19IL2/L19TNF have been observed in patients with injectable melanoma lesions of stage III or IV, for injected and non-injected lesions.

The proposed clinical phase II study plans to investigate the intralesional administration of 6.5 Mio IU of L19IL2 (~1.08 mg) and 200 µg of L19TNF to be administered in an approximate volume of 1.0 mL as a single or multiple intratumoral injections in patients with high-risk BCC or cSCC.

There is a high medical need for non-invasive therapeutic strategies with a comparable good response rate and high recurrence free survival for treatment of patients with BCC or cSCC, who cannot be treated by or refuse surgery. Surgery is not always applicable, as it may not be feasible due to the anatomic location, may have a poor cosmetic outcome for the patient or is generally not accepted as treatment strategy by the patient. However, current non-surgical treatment strategies have a considerably reduced response rate and recurrence free survival. Based on the favorable results for injected and non-injected lesions obtained in the phase II study of L19IL2/L19TNF and the good safety profile seen in the subsequent phase III study, both in stage III or IV melanoma patients, we believe, that patients with BCC or cSCC will profit from intralesional treatment with L19IL2/L19TNF.

ELIGIBILITY:
Inclusion Criteria:

* High-risk, localized (non-metastatic, node negative, single or multifocal) BCC or cSCC amenable to intratumoral injection.
* Patients with injectable and measurable regional cutaneous or subcutaneous in-transit or satellite metastasis but without regional nodal involvement are also eligible.
* Male or female patients, age 18 - 100 years.
* ECOG Performance Status/WHO Performance Status ≤ 1.
* Hemoglobin > 10.0 g/dL.
* Platelets > 100 x 10^9/L.
* ALT and AST, GGT and Lipase ≤ 1.5 x the upper limit of normal (ULN).
* Serum creatinine < 1.5 x ULN and GFR > 60 mL/min.
* All acute toxic effects (excluding alopecia) of any prior therapy must have resolved to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE v. 5.0) Grade ≤ 1 unless otherwise specified.
* Women of childbearing potential (WOCBP) must have negative pregnancy test results at screening. WOCBP must be using, from screening to three months following the last study drug administration, highly effective contraception methods, as defined by the "Recommendations for contraception and pregnancy testing in clinical trials" issued by the Head of Medicine Agencies' Clinical Trial Facilitation Group and which include, for instance, progesterone-only or combined (estrogen- and progesterone-containing) hormonal contraception associated with inhibition of ovulation, intrauterine devices, intrauterine hormone-releasing systems, bilateral tubal occlusion, vasectomised partner.
* Male patients with WOCBP partners must agree to use simultaneously two acceptable methods of contraception (i.e. spermicidal gel plus condom) from the screening to three months following the last study drug administration.
* Willingness and ability to comply with the scheduled visits, treatment plan, laboratory tests and other study procedures.

Exclusion Criteria:

* Previous or concurrent cancer type that is distinct from the cancers being evaluated in this study, except any cancer curatively treated more than 2 years prior to study entry.
* Patients may have previously received topical or systemic chemotherapy, immunotherapy or radiation therapy on the tumor sites. Such therapies must be completed at least 4 weeks prior to study drug administration.
* Patients with node positive BCC/cSCC who are candidate to SHH inhibitor or checkpoint inhibitor therapy.
* Presence of active severe bacterial or viral infections or other severe concurrent disease, which, in the opinion of the investigator, would place the patient at undue risk or interfere with the study. In particular a documented test for HIV, HBV and HCV excluding active infection is needed.
* History within the last year of acute or subacute coronary syndromes including myocardial infarction, unstable or severe stable angina pectoris, inadequately treated cardiac arrhythmias and heart insufficiency (any grade, New York Heart Association (NYHA) criteria).
* Any abnormalities observed during baseline ECG investigations that are considered clinically significant by the investigator.
* Known arterial aneurysms.
* INR > 3.
* Uncontrolled hypertension.
* Known uncontrolled coagulopathy or bleeding disorder.
* Known hepatic cirrhosis or severe pre-existing hepatic impairment.
* Moderate to severe respiratory failure.
* Active autoimmune disease.
* Patient requires or is taking systemic corticosteroids (>5 mg/day) or other immunosuppressant drugs on a long-term basis. Limited use of corticosteroids to treat or prevent acute hypersensitivity reactions and asthma/COPD is not considered an exclusion criterion.
* Known history of allergy to IL2, TNF, or other human proteins/peptides/antibodies.
* Pregnancy or breast-feeding.
* Ischemic peripheral vascular disease (Grade IIb-IV).
* Severe diabetic retinopathy.
* Recovery from major trauma including surgery within 4 weeks prior to enrollment.
* Solid organ transplant recipient or patient with iatrogenic or pathologic severe immune suppression.
* Any conditions that in the opinion of the investigator could hamper compliance with the study protocol.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-09-02 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Efficacy of L19IL2/L19TNF in CR | Tumor Assessment/Safety visit (Week 6, Day 36)
  Objective Response Rate (Complete Response CR) for each tumor type from beginning of treatment according to RECIST v1.1 criteria.
Efficacy of L19IL2/L19TNF in PR | Tumor Assessment/Safety visit (Week 6, Day 36)
  Objective Response Rate (Partial Response PR) for each tumor type from beginning of treatment according to RECIST v1.1 criteria.

SECONDARY OUTCOMES:
Pathological Response | At Surgery
  Efficacy of L19IL2/L19TNF measured as Pathological Response for each tumor type at the time of surgery.
Safety (AE) | Throughout study completion for each patient, an average of 12 weeks for each patient
  Safety of intratumoral administration of L19IL2/L19TNF, assessed by Common Toxicity Criteria (version 5.0, CTCAE)
Safety: ECG | Before first drug administration at Day 1 and at the Tumor Assessment Visit at Day 36 (Week 6).
  Electrocardiogram (ECG) findings. In particular, data about QT/QTc intervals will be collected and analysed for QT/QTc prolongation potentially caused by treatment
Safety: change in vital signs | Before first drug administration at Day 1, Day 8, Day 15, Day 22 and at the Tumor Assessment Visit at Day 36 (Week 6).
  Measurement of heart rate (beats per minute)
Safety: change in vital signs | Before first drug administration at Day 1, Day 8, Day 15, Day 22 and at the Tumor Assessment Visit at Day 36 (Week 6).
  Measurement of blood pressure (mmHg)

CONTACTS AND LOCATIONS:
Locations (11):
- Germany (8):
  - Universitätsklinikum Augsburg, Augsburg
  - Charité Universitätsmedizin Berlin, Berlin
  - University Hospital Carl Gustav Carus, Dresden
  - Universitätsklinikum Essen (AöR), Essen
  - Nationales Centrum für Tumorerkrankungen (NCT), Heidelberg
  - University Medical Center Schleswig Holstein, Kiel
  - Universitätsklinikum Regensburg, Regensburg
  - Tübingen University Hospital, Tübingen
- Centrum Onkologii-Instytut im. Marii Skłodowskiej-Curie Warszawa, Warsaw, Poland
- Switzerland (2):
  - Kantonsspital St.Gallen, Clinical Trials Unit, Dermatologie und Venerologie, Sankt Gallen
  - Universitätsspital Zürich (USZ), Zurich

IPD SHARING:
Plan to Share IPD: No